CLINICAL TRIAL: NCT06400602
Title: Integrative Health Coaching for Back Pain: An Emergency Department-to-Home Recovery Model
Brief Title: Health Coaching for Back Pain After Emergency Department Discharge
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Rogelio Coronado, Research Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 231665
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual ED Care plus Health Coaching (Experimental)
  Interventions: Behavioral: Usual ED Care plus Health Coaching
- Usual ED Care plus Education (Active Comparator)
  Interventions: Behavioral: Usual ED Care plus Education

INTERVENTIONS:
Behavioral: Usual ED Care plus Health Coaching — Patients will participate in eight remotely-delivered sessions of health coaching after ED discharge. Patients will receive usual care during their ED visit.
  Arms: Usual ED Care plus Health Coaching
Behavioral: Usual ED Care plus Education — Patients will participate in eight remotely-delivered sessions of education after ED discharge. Patients will receive usual care during their ED visit.
  Arms: Usual ED Care plus Education

SUMMARY:
The goal of this two-group randomized trial is to determine the feasibility and acceptability of a remotely-delivered health coaching intervention offered in conjunction with usual care for patients with an acute exacerbation of chronic low back pain who present to the emergency department (ED).

The main questions this feasibility trial aims to answer are:

* Is our health coaching intervention and randomized trial methodology feasible to conduct?
* Is our health coaching intervention acceptable to participants and ED providers?

Participants will be randomized to one of two groups (usual ED care plus health coaching or usual ED care plus education) and complete outcome assessments at 3 and 6 months after ED discharge. Participants and ED providers will also complete an interview.

DETAILED DESCRIPTION:
This study is a two-group randomized feasibility trial of usual ED care plus either remote health coaching or remote education in patients with acute exacerbation of chronic low back pain presenting to the ED. We hypothesize that our health coaching intervention and randomized trial methodology will be feasible and that our health coaching intervention will be acceptable to participants and ED providers.

Forty participants will be randomized (20 per group), with 36 (90%) retained in the trial up to 6 months follow-up. Eligible patients presenting to the ED with a chief complaint of acute exacerbation of chronic low back pain will be randomized. Patients will be enrolled during or shortly after their ED visit, asked to complete a baseline questionnaire, and then randomized. Randomized participants will receive 8 calls from either a health coach or education provider, and be asked to complete assessments at 3 and 6 months after ED discharge. Interviews will be conducted with randomized participants and 15 ED providers asking about their experience with the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Chief complaint of musculoskeletal LBP
2. Meets NIH-supported chronic LBP criterion (e.g., pain greater than 3 months that has resulted in pain on at least half the days in the past 6 months)
3. Age 18 years of age or older
4. English-speaking

Exclusion Criteria:

1. Requires hospitalization for an acute medical condition or active comorbidity
2. In the opinion of the investigator has a severe psychiatric or behavioral diagnosis or substance use disorder that would interfere with the ability to perform the intervention and complete follow-up
3. Involved in litigation related to the LBP condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility - study enrollment | Baseline
  Percentage of eligible patients enrolled into study
Feasibility - study retention | 3 and 6 months after ED discharge
  Percentage of enrolled participants who complete assessments
Feasibility - session attendance | 3 months after ED discharge
  Median and range of sessions attended
Feasibility - Feasibility of Intervention Measure (FIM) | 3 months after ED discharge
  4-item questionnaire assessing feasibility of an intervention. Averaged scores range from 1 to 5, with higher scores indicating greater feasibility.
Acceptability - Acceptability of Intervention Measure (AIM) | 3 months after ED discharge
  4-item questionnaire assessing acceptability of an intervention. Averaged scores range from 1 to 5, with higher scores indicating greater acceptability.
Acceptability - Intervention Appropriateness Measure (IAM) | 3 months after ED discharge
  4-item questionnaire assessing appropriateness of an intervention. Averaged scores range from 1 to 5, with higher scores indicating greater appropriateness.
Perceptions of intervention | 3 months after ED discharge
  Perceptions of intervention as assessed through an interview

SECONDARY OUTCOMES:
Disability - Oswestry Disability Index | Baseline, 3 months after ED discharge, 6 months after ED discharge
  10-item questionnaire assessing back-related disability. Scores range from 0 to 100, with higher scores indicating higher disability.
Physical Function - Patient-Reported Outcomes Measurement Information System (PROMIS) | Baseline, 3 months after ED discharge, 6 months after ED discharge
  4-item PROMIS questionnaire assessing physical function. Scores are reported as t-scores, with higher scores indicating higher physical function.
Pain Interference - Patient-Reported Outcomes Measurement Information System | Baseline, 3 months after ED discharge, 6 months after ED discharge
  4-item PROMIS questionnaire assessing pain interference. Scores are reported as t-scores, with higher scores indicating higher pain interference.
Pain Intensity - Patient-Reported Outcomes Measurement Information System | Baseline, 3 months after ED discharge, 6 months after ED discharge
  Single item question assessing level of pain intensity. Scores range from 0 to 10, with higher scores indicating higher pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Rogelio Coronado, PT, PhD, Principal Investigator — Vanderbilt University Medical Center; Kristin Archer, PhD, DPT, Study Director — Vanderbilt University Medical Center; Sean Collins, MD, Study Director — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Tennessee Valley Healthcare System - Nashville VA Medical Center, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No